CLINICAL TRIAL: NCT03753841
Title: Flexible Endoscopic Evaluation of Swallowing (FEES) to Determine Neurological Patients' Oral Diet
Brief Title: FEES to Determine Neurological Intensive Care Patients' Oral Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Tobias Braun, Principal Investigator, University of Giessen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI 208/16-1
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Dysphagia; Aspiration Pneumonia; Deglutition Disorders; Intensive Care Neurological Disorder
Keywords: Dysphagia; Aspiration; Management of Dysphagia; Deglutition Disorders; Deglutition; FEES; Intensive Care Neurological Disorder
MeSH Terms: conditions — Deglutition Disorders; Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustment of oral diet (Active Comparator): Patients who need a change in their diet regime, in whom FEES shows that they have not the adequat diet.
  Interventions: Other: Adjustment of oral diet
- No adjustment of oral diet (No Intervention): Patients who have the adequat diet based on FEES findings.

INTERVENTIONS:
Other: Adjustment of oral diet — Adjustment of oral diet based on findings in fiberendoscopic evaluation of swallowing (FEES)
  Arms: Adjustment of oral diet

SUMMARY:
Dysphagia is associated with high rates of mortality and morbidity. Adjusting the oral diet of ICU-patients based on flexible endoscopic evaluation of swallowing (FEES) findings might reduce pneumonia rate, mortality and need for intubation/tracheotomy.

DETAILED DESCRIPTION:
Dysphagia, a common complication in neurological disorders, leads to high rates of mortality and morbidity. It is prevalent in critically ill patients, especially those who need mechanical ventilation. The investigators therefore investigate the effect of adjusting the oral diet of our intensive care unit (ICU) patients based on flexible endoscopic evaluation of swallowing (FEES) findings, thereby assessing the impact of FEES on a neurological ICU. All patients treated on the investigators neurological ICU will be eligible for this study.

The investigators will correlate findings with baseline data, disability status, pneumonia and duration of hospitalisation, as well as a need for mechanical ventilation or a tracheotomy.

ELIGIBILITY:
Inclusion Criteria:

* Treatment on neurological ICU
* Clinical suspicion of Dysphagia

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Pneumonia Rate | Up to 130 days
  self-explanatory
Mortality | Up to 130 days
  self-explanatory

SECONDARY OUTCOMES:
Length of stay in hospital | Up to 130 days
  self-explanatory
Intubation/Tracheotomy | Up to 130 days
  Rate of Intubation/Tracheotomy

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Braun, M.D., Principal Investigator — University of Giessen
Locations (1):
- Universitätsklinikum Gießen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
The authors declare that the data supporting the findings of this study will be available within the published article(s). The data that support the findings of this study will not be publically available due to local medical data protection policies.